CLINICAL TRIAL: NCT00851409
Title: An Open-label Exploratory Phase II Study of the Safety and Immunogenicity of Repeated "rhC1INH" Administration of 50 U/Kg in Patients With Hereditary C1 Inhibitor Deficiency ("HAE")
Brief Title: A Study of the Safety and Immunogenicity of Repeated rhC1INH Administration
Acronym: OPERA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharming Technologies B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1 1207
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Results first posted 2013-01-31 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-04

CONDITIONS: Genetic Disorders; Hereditary Angioedema
MeSH Terms: conditions — Genetic Diseases, Inborn; Angioedemas, Hereditary | interventions — Complement C1 Inhibitor Protein; conestat alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Recombinant Human C1 Inhibitor (Other): Weekly administration of 50 IU/kg Recombinant Human C1 Inhibitor
  Interventions: Drug: Recombinant Human C1 Inhibitor

INTERVENTIONS:
Drug: Recombinant Human C1 Inhibitor — 50 IU/kg "rhC1INH", "IV" injection over 4 to 5 minutes, once weekly over an 8-week treatment period.
  Other Names: "rhC1INH"; Ruconest

SUMMARY:
Hereditary angioedema ("HAE") is a disease characterized by recurrent tissue swelling affecting various body locations. Recent literature shows that patients with frequent attacks may benefit from long-term prophylaxis. This study aims to evaluate the safety and prophylactic effect of weekly administrations of 50 IU/kg recombinant C1 Inhibitor ("rhC1INH").

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years
* Signed informed consent
* Comfirmed diagnosis of HAE with baseline plasma level of functional C1INH activity of less than 50% of normal, and/or proven HAE ,mutation in C1INH gene.

Exclusion Criteria:

* A history of anaphylaxis or severe allergy (i.e. requiring medication) to food, proteins and/or drugs.
* A history of allergic reactions to C1INH products or rabbit protein.
* Any reported SAE related to study drug administration (withdrawal criterium)
* Elevated IgE against rabbit dander (>0.35 kU/L; ImmunoCap assay; Phadia)
* A diagnosis of acquired C1INH deficiency.
* Woman of child bearing potential, pregnancy or breast-feeding
* previous treatment within the last 3 months with plasma-derived C1INH
* Any clinically significant abnormality in the routine haematology, biochemistry and urinalysis
* Any condition or treatment that in the opinion of the investigator might interfere with the evaluation of the study objectives.
* Any changes since screening that would exclude subject based on above exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-06; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Giannetti, MD, Study Chair — COO Pharming
Locations (2):
- For information on sites, please contact Pharming Technologies, Leiden, Netherlands
- Emergency County Hospital, Internal Medicin Clinica, Allergology-Immunology Department, Târgu Mureş, Romania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with a history of frequent attacks, defined as "HAE" attacks occurring at least every two weeks were included in the study.
Groups:
- Recombinant Human C1 Inhibitor: Weekly administration of 50 IU/kg recombinant human C1 inhibitor
  Recombinant Human C1 Inhibitor : 50 IU/kg "rhC1INH", "IV" injection over 4 to 5 minutes, once weekly over an 8-week treatment period.
Period: Overall Study
Arm/Group | Recombinant Human C1 Inhibitor
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Recombinant Human C1 Inhibitor
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: HAE Attacks/Week
Description: Prior to the treatment period, patients enrolled in the study, were asked about the amount of "HAE" attacks in the past 2 years, (calculated to attacks/week), this number is defined as "Historical". During the treatment period, patients received a dose of 50 IU/kg of "rhC1INH" administered by slow "IV" injection over 4 to 5 minutes, once a week during an eight week period. The amount of attacks during this period is defined as "Prophylaxis" (calculated to attacks/week).
Time Frame: 8 weeks
Measure: Mean (95% Confidence Interval); unit: attacks/week
Groups:
- Recombinant Human C1 Inhibitor: Recombinant Human C1 Inhibitor : 50 IU/kg "rhC1INH", "IV" injection over 4 to 5 minutes, once weekly over an 8-week treatment period.
Arm/Group | Recombinant Human C1 Inhibitor
Number analyzed (Participants) | 25
attacks/week
  Historical | 0.9 [0.51 to 1.30]
  Prophylaxis | 0.4 [0.27 to 0.56]

2. Secondary Outcome: The Evaluation of Pharmacokinetic/ Pharmacodynamic ("PK/PD")Parameters.
Description: "PK/PD" parameters will be based on concentration time curves after the 1st and 8th "rhC1INH" administration.(ratio visit 8/ visit 1, based on the area under the curve from baseline up to 4 hours after administration (AUC 0-4)
Time Frame: 8 weeks
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Recombinant Human C1 Inhibitor
Number analyzed (Participants) | 25
ratio
  Functional C1 Inhibitor level | 1.06 [0.98 to 1.14]
  Antigenic C1 Inhibitor level | 1.02 [0.91 to 1.15]
  C4 level | 1.00 [0.74 to 1.33]

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events ("TEAEs") were defined as events with start from onset of study drug administration. All Serious Adverse Events("SAEs")are listed.
Description: All Adverse Events ("AEs")occurring within 7 days of onset after study drug administration have been listed.
Arm/Group | Recombinant Human C1 Inhibitor
Serious Adverse Events (participants affected / at risk) | 2/25
Other Adverse Events (participants affected / at risk) | 2/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Human C1 Inhibitor (N=25)
Appendicitis (Infections and infestations) | 1 (1)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Human C1 Inhibitor (N=25)
Anaemia-mild (Blood and lymphatic system disorders) | 1 (1)
Anaemia-moderate (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator must provide a copy of any results communication to the sponsor for review at least 30 days prior to its submission or disclosure. The sponsor may request to delete information identified by sponsor as confidential information prior to submitting such manuscript and/or abstract for publication. For a multi-center study, the investigator must wait (i) at least 24 months after the study is completed at all sites or (ii) until after the multi-center publication.